CLINICAL TRIAL: NCT03302260
Title: IMPROVE (Identifying Methods for Postpartum Reduction of Vascular Events): Pilot Randomized Controlled Trial
Brief Title: Identifying Methods for Postpartum Reduction of Vascular Events: Pilot Randomized Controlled Trial
Acronym: IMPROVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB17-1264
Record Dates: First submitted 2017-09-20; First posted 2017-10-05 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pre-Eclampsia
Keywords: maternal health; pregnancy; pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The nature of the intervention (i.e., the CardioPrevent® cognitive-behavioural lifestyle counsellor) does not lend itself to blinding of the participant. However, the research assistant responsible for the outcome assessments will be blinded to each participant's group allocation and will be instructed not to ask any questions pertaining to the study intervention. The study statistician will also be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control arm will receive standard postpartum clinical care through the participants' usual healthcare providers. No intervention will be administered. Participants in both arms will receive educational material about the risk of CVD, and CVD prevention for women with HDP from the Preeclampsia Foundation.
- CardioPrevent® Program (Experimental): In addition to standard care, participants randomized to the intervention arm will also receive the CardioPrevent® Program. This is a 1-year, evidence-based behaviour change lifestyle program that consists of 25 contacts (in person, by phone and in groups) with a trained lifestyle counsellor to facilitate desired lifestyle behaviours within the participants' own social context. Participants in both arms will receive educational material about the risk of CVD, and CVD prevention for women with HDP from the Preeclampsia Foundation.
  Interventions: Behavioral: CardioPrevent® Program

INTERVENTIONS:
Behavioral: CardioPrevent® Program — This is a 1-year, evidence-based behaviour change lifestyle program that consists of 25 contacts (in person, by phone and in groups) with a trained lifestyle counsellor to facilitate desired lifestyle behaviours within the participants' own social context.
  Arms: CardioPrevent® Program

SUMMARY:
IMPROVE is a pilot RCT with a behavioral intervention component (CardioPrevent program). The primary objectives of this pilot study are to assess the feasibility of the implementation of a postpartum CVD prevention lifestyle program in women with a HDP as well as the transferability and fidelity of the Ottawa-based CardioPrevent® program to a centre in Calgary (following a "Train the Trainer" model). Secondary objectives include an initial evaluation of the effectiveness of this intervention on clinical outcomes and measures of microvascular function between study arms at one year.

DETAILED DESCRIPTION:
1. Background and Rationale

   Cardiovascular disease (CVD) (i.e., coronary artery disease, stroke, and peripheral arterial disease) is one of the leading causes of morbidity and mortality in Canada, particularly amongst women. Women with hypertensive disorders of pregnancy (HDP) represent one of the highest-risk populations for premature CVD and CVD mortality. The 2011 American Heart Association (AHA) Guidelines on the prevention of CVD in women now include HDP as an independent CVD risk factor in the evaluation of CVD risk. To achieve "ideal cardiovascular health" targets, healthy lifestyle modifications are suggested as first-line therapy, with pharmacotherapy as second line. The immediate postpartum period may be an early window of opportunity for early upstream CVD prevention, capitalizing on a woman's increased motivation to improve her health. Despite these recommendations and opportunity for early CVD prevention, there is little published data, and, in particular, there are no randomized controlled trials (RCT) assessing the short-term or long-term effectiveness of lifestyle interventions in women with HDP.

   To address this important clinical problem and knowledge gap, the interdisciplinary IMPROVE team adapted the evidence-based University of Ottawa Heart Institute CardioPrevent® Lifestyle program to proactively address the unique barriers to, and facilitators of behaviour change in early postpartum women with HDP. Prior to undertaking a widespread evaluation of CardioPrevent® in a CVD prevention study for women with HDP, a pre-assessment of the feasibility of this postpartum lifestyle program using this research approach through a pilot study is essential. In addition, this pilot study will provide important information on CardioPrevent®'s effectiveness on modifying clinically-important cardiovascular-related clinical outcomes and novel, non-invasive measures of microvascular function in early postpartum women with HDP to inform the design of a larger CVD prevention study. This pilot RCT will be the first to assess the feasibility and effects of a one-year postpartum-specific CVD prevention lifestyle program in women with a HDP.
2. Research Questions & Objectives

   The primary objectives of this pilot study are to assess the feasibility of the implementation of a postpartum CVD prevention lifestyle program in women with a HDP as well as the transferability and fidelity of the Ottawa-based CardioPrevent® program to a centre in Calgary (following a "Train the Trainer" model). Secondary objectives include: an initial evaluation of the effectiveness of this intervention on clinical outcomes and measures of microvascular function between study arms at one year.
3. Methods

Study Design: A 2-year, single centre, single-blind, pilot randomized controlled trial (RCT).

Study Population (Inclusion/Exclusion Criteria): Women with a HDP (i.e., preeclampsia, eclampsia or gestational hypertension) delivering at the Foothills Medical Centre will be invited to participate. Women with pre-existing chronic hypertension, diabetes (type 1 or type 2), kidney disease or cardiovascular disease (coronary artery, cerebrovascular and peripheral arterial) will be excluded.

Intervention: CardioPrevent® Program - a one year, evidence-based cardiovascular prevention program that consists of 25 contacts (either in person or by phone) with a trained behaviour change counsellor to facilitate desired lifestyle behaviours within the participants' own social context.

Control: Standard clinical postpartum care. All Participants: Participants in both arms will receive educational material about the risk of CVD and CVD prevention for women with HDP from the Preeclampsia Foundation.

Sample size: A total of 84 women will be recruited (42 in each arm). Recruitment & Retention: There are over 7000 deliveries per year at the FMC. Using a conservative estimate of 7% prevalence of HDP (as it is a tertiary care referral centre), approximately 245 women (10 per week) will have HDP over our 6-month recruitment period. The investigators anticipate recruiting 2-3 eligible women per week to reach the target sample size in 6 months. To minimize loss to follow-up, they plan to use participant incentives such as covering the costs of parking and childcare.

ELIGIBILITY:
Inclusion Criteria:

* adult women aged 18 years or older;
* diagnosis of a HDP (i.e., preeclampsia, eclampsia or gestational hypertension);
* delivering at The Foothills Medical Centre (FMC) in Calgary, Alberta;
* ability to read, write, understand, and provide informed consent in English; and
* have telephone access.

Exclusion Criteria:

* pre-existing vascular disease (coronary artery disease [i.e., stable angina, unstable angina,
* myocardial infarction, percutaneous coronary intervention or coronary artery bypass surgery],
* cerebrovascular disease [i.e., ischemic stroke or transient ischemic attack], or peripheral arterial
* disease [i.e., known abnormal ankle-brachial indices, symptoms of intermittent claudication, or
* bypass surgery to the extremities]);
* chronic hypertension;
* diabetes (type 1 or type 2);
* pre-pregnancy kidney disease;
* planning another pregnancy within one year;
* counselling may not be appropriate (i.e., impaired cognition);
* live more than 200 km outside the Calgary region; and
* planning to move outside the Calgary region within one year of randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Study feasibility - recruitment | 2 years
  Acceptance of the study by women with HDP (i.e., feasibility) measured by recruitment rate of ≥ 20% over a 6-month time period (as per weekly recruitment logs).
Study feasibility - adherence | 2 years
  Acceptance of the study by women with HDP (i.e., feasibility) measured by participant adherence of ≥ 80% to the lifestyle program (i.e., 20/25 contacts with counsellor completed).
Study feasibility - study completion | 2 years
  Acceptance of the study by women with HDP (i.e., feasibility) measured by overall study completion rate of ≥ 75% of participants.
Study feasibility - participant satisfaction | 2 years
  Acceptance of the study by women with HDP (i.e., feasibility) measured by participant satisfaction score of ≥ fair on the Client Satisfaction Questionnaire at the end of study.
Implementation and fidelity of CardioPrevent® at the University of Calgary (a second centre) - audits | 2 years
  Implementation and fidelity of CardioPrevent® at the University of Calgary (a second centre) measured by standardized audits.
Implementation and fidelity of CardioPrevent® at the University of Calgary (a second centre) - clinical outcomes | 2 years
  Implementation and fidelity of CardioPrevent® at the University of Calgary (a second centre) measured by similar clinical outcomes between sites.

SECONDARY OUTCOMES:
Weight | 2 years
  Comparison of weight (kg) between both study arms at one year of follow-up.
Body mass index (BMI) | 2 years
  Comparison of BMI (kg/m^2) between both study arms at one year of follow-up.
Waist-to-hip ratio | 2 years
  Comparison of waist-to-hip ratio between both study arms at one year of follow-up .
Smoking status | 2 years
  Comparison of smoking status between both study arms at one year of follow-up (CO levels <10ppm confirmatory for non-smoking).
Postpartum depression | 2 years
  Comparison of postpartum depression between both study arms at one year of follow-up (measured by the Edinburgh Postnatal Depression Scale).
Blood pressure | 2 years
  Comparison of blood pressure (mmHg) between both study arms at one year of follow-up.
Fasting lipids | 2 years
  Comparison of fasting lipids (mmol/L) between both study arms at one year of follow-up.
Fasting glucose | 2 years
  Comparison of fasting glucose (mmol/L) between both study arms at one year of follow-up.
HbA1C | 2 years
  Comparison of HbA1C (%) between both study arms at one year of follow-up.
Urine albumin to creatinine ratio | 2 years
  Comparison of urine albumin to creatinine ratio between both study arms at one year of follow-up.
Metabolic syndrome | 2 years
  Comparison of metabolic syndrome between both study arms at one year of follow-up measured by z-score (calculated using Adult Treatment Panel (ATP) III Criteria for Metabolic Syndrome).
CVD risk | 2 years
  Comparison of CVD risk between both study arms at one year of follow-up.
Microvascular function - flow mediated dilation (FMD) | 2 years
  Comparison of FMD between both study arms at one year of follow-up.
Microvascular function - brachial artery hyperemic velocity | 2 years
  Comparison of brachial artery hyperemic velocity between both study arms at one year of follow-up.
Microvascular function - peripheral arterial tonometry (PAT) | 2 years
  Comparison of PAT between both study arms at one year of follow-up.
Changes in amount of physical activity recorded in questionnaire | 2 years
  Comparison of amount of physical activity (IPAQ short form) logs between both study arms at one year of follow-up.
Changes in amount of physical activity recorded in activity logs | 2 years
  Comparison of amount of physical activity (physical activity logs) logs between both study arms at one year of follow-up.
Changes in amount of physical activity captured by accelerometer | 2 years
  Comparison of amount of physical activity (accelerometer data) between both study arms at one year of follow-up.
Changes in dietary behavior | 2 years
  Comparison of eating behaviors (Rapid eating assessment of patients) questionnaire between both study arms at one year of follow-up.
Changes in nutrient status | 2 years
  Comparison of nutrient status (measured by three days of prospective food logs) between both study arms at one year of follow-up.

IPD SHARING:
Plan to Share IPD: No